CLINICAL TRIAL: NCT05340348
Title: Formation of a Patientheque in Patients With a Beginner Psychosis .
Brief Title: Patientheque in Patients With a Psychosis .
Acronym: LONGIPEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC20.0097
Record Dates: First submitted 2022-03-08; First posted 2022-04-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia Prodromal; Schizophrenia, Childhood; Schizophrenia
Keywords: Schizophrenia; Patient library
MeSH Terms: conditions — Schizotypal Personality Disorder; Schizophrenia, Childhood; Schizophrenia | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Monocentric interventional study with minimal risks and constraints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient library (Other): All the patients are included in one arm. They will undergo various type of samples.
  Interventions: Other: Blood samples (36 mL) + fecal samples + hair sample

INTERVENTIONS:
Other: Blood samples (36 mL) + fecal samples + hair sample — Blood samples at inclusion, 2 years later and/or if relapse, fecal samples at inclusion and every years for 5 years, hair sample at inclusion
  Other Names: Patient library

SUMMARY:
Establishment of a patient library for patients who have had a first psychotic episode and who have an "at risk" status for psychotic disorder (GRD, APS, BLIPS group) or a psychosis threshold during CAARMS administration. Samples are taken on inclusion, at 2 years, and if relapse or significant clinical event within 5 years of inclusion, on 250 patients for 10 years.

DETAILED DESCRIPTION:
The constitution of this patient library will include results of clinical tests carried out in current practice, neurocognitive tests, blood samples, audio recordings, clinical follow-up, urine samples, fecal samples, brain imaging, EEG.

ELIGIBILITY:
Inclusion Criteria:

* Major and or minor aged 15 to 30 assessed within the CEVUP (Consultation for the Assessment of Psychological Vulnerability) and cared for at the psychiatry center as part of a first psychotic episode (Diagnosis CIM 10: F20 -F29 first hospitalization). These patients are referred by care and medico-social partners (general practitioners, school doctors, school nurses, educators, addictologists, psychiatrists
* "At risk" status for psychotic disorder (GRD, APS, BLIPS group) or psychosis threshold during the CAARMS test (psychometric scale for the assessment of psychotic symptoms)
* Consent of the patient or his legal guardian

Exclusion Criteria:

* History of psychosis for more than one year
* "Not at risk" status for psychotic disorder on the CAARMS (psychometric scale for the assessment of psychotic symptomatology)
* IQ<70 (WAIS)
* Neurological disorder or other health problem that may explain the disorders
* Refusal to participate - History of psychosis for more than one year

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2027-07-25 (Estimated); Study Completion 2032-07-25 (Estimated)

PRIMARY OUTCOMES:
CAARMS (Comprehensive assessment of at-risk mental states) score. | 5 years
  The test will determine the mental state of the patient :
  * "Not at risk of psychosis"
  * "At risk of psychosis"
  * "Psychosis threshold exceeded"
  It is organized into 7 clinical dimensions: 1) positive symptoms 2) cognitive changes: attention / concentration 3) emotional disturbance 4) negative symptoms 5) behavioral change 6) physical and motor changes 7) general psychopathology.
  Each category is scored between 0 and 6 depending on the level of intensity, frequency and duration of each symptom.
  In order to determine if a subject meets the UHR criteria for CAARMS, only the first category (positive symptoms) and its four subscales are used according to a scoring algorithm.

SECONDARY OUTCOMES:
CAARMS sub-assemblies | 5 years
  If the patient is classified at risk of psychosis, the test will classify this risk into one of the three following categories : trait and state risk factor group, APS (attenuated psychotic symptoms) group, BLIPS (Brief, Limited or Intermittent Psychotic Symptoms) group.

CONTACTS AND LOCATIONS:
Overall Officials: Michel WALTER, Principal Investigator — CHRU BREST
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital (UH). Requestors will be required to sign and complete a data access agreement.